CLINICAL TRIAL: NCT05316922
Title: Protection From Iatrogenic Hypothyroidism Patients With MBL and Pediatric Patients With HL and Non-HL Needing Radiotherapy on Thyroid Site
Brief Title: TSH Suppression During Radiotherapy on Thyroid Site to Prevent Iatrogenic Hypothyroidism in Pediatric Cancer Patients
Acronym: WIN-HYPO2021
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INT122/21
Record Dates: First submitted 2021-09-14; First posted 2022-04-07 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Hypothyroidism; Irradiation
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine; Antithyroid Agents

STUDY DESIGN:
Intervention Model Description: Prospective, non-blinded, randomised two cohorts study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TSH suppression during irradiation (Experimental): From 14 days beforehand and throughout their RT, patients in the experimental arm will receive L-thyroxine in the morning, starting with 1-2 μg/kg, and adjusting the dose every 3 days to ensure TSH < 0.3 μIU/mL before RT beginning. The 0.3 μIU/mL threshold is just below normal range not causing hyperthyroidism, and is defined as "mild" TSH suppression. Based on hormone status, L-thyroxine doses will be gradually increased to patients' individual minimum TSH-suppressive dose before starting RT, maintained throughout the treatment, then rapidly tapered off and stopped. During radiation treatment course will be checked twice a week for serum FT3, FT4, TSH assays in order to maintain TSH < 0.3 μIU/mL, possibly without exceeding normal levels of FT3 and FT4. Once a week patients will also have a full visit and any other blood examination according to protocol in use and Institutional practice.
  Interventions: Drug: Levothyroxine
- Any TSH suppression during irradiation (No Intervention): Patient in the standard arm will perform radiotherapy treatment without any TSH suppression. At the end of radiation they will do serum FT3, FT4, TSH assay and then, after one year from RT, thyroid ultrasound + serum FT3, FT4, TSH assay.

INTERVENTIONS:
Drug: Levothyroxine — Levothyroxine is used to treat hypothyroidism (low thyroid function). This medicine is given when your thyroid does not produce enough of this hormone on its own.
  Other Names: Thyroid drugs
  Arms: TSH suppression during irradiation

SUMMARY:
To offer the possibility of a treatment that could achieve a meaningful reduction in the incidence of post-radiation therapy hypothyroidism. Thyroid dysfunction may develop from a few months to several years after patients have completed their radiation treatment. In children with chronic diseases, or given lengthy anti-neoplastic treatments, recurrent or persistent endocrine disorders may have a negative effect on growth and development into adulthood.

DETAILED DESCRIPTION:
Patients will undergo basal thyroid ultrasound and FT3, FT4, TSH assay. Simulations with computed tomography, and computer assisted three-dimensional treatment planning with a dose volume histogram will be used to identify thyroid volumes and corresponding RT isodose distributions.

The enrolled patients will be randomly assigned (1:1) to TSH suppression group (experimental group) or non-TSH suppression group (control group). Random allocation will be managed centrally by Clinical epidemiology and Trial organization of the Fondazione IRCCS Istituto Nazionale dei Tumori. The randomization list will be generated by SAS software. Investigators and patients will not be masked to treatment allocation.

From 14 days beforehand and throughout their RT, patients in the experimental arm will receive L-thyroxine in the morning on an empty stomach (half an hour before breakfast), starting with 1-2 μg/kg, and adjusting the dose every 3 days to ensure TSH < 0.3 μIU/mL before RT beginning. The 0.3 μIU/mL threshold is just below normal range not causing hyperthyroidism, and is defined as "mild" TSH suppression. Based on hormone status, L-thyroxine doses will be gradually increased to patients' individual minimum TSH-suppressive dose before starting RT, maintained throughout the treatment, then rapidly tapered off (half dose the next day after RT, 25% the following day and stop).

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with medulloblastoma, Hodgkin/non-Hodgkin Lymphoma before radiotherapy (RT) planning including thyroid parenchyma without previous primary or secondary hypothyroidism;
2. Written informed consent prior to any study-specific analysis and/or data collection.

Exclusion Criteria:

1. Any patient with medulloblastoma, Hodgkin/non-Hodgkin Lymphoma after radiotherapy including thyroid parenchyma;
2. Not signed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Hypothyroidism-free survival | 3 years
  Hypothyroidism-free survival at 3 years after radiotherapy including part or the whole thyroid parenchyma on the intention-to-treat population will be the main end-point.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prpic M, Kruljac I, Kust D, Suton P, Purgar N, Bilos LK, Gregov M, Mrcela I, Franceschi M, Djakovic N, Frobe A. Dose-volume derived nomogram as a reliable predictor of radiotherapy-induced hypothyroidism in head and neck cancer patients. Radiol Oncol. 2019 Nov 20;53(4):488-496. doi: 10.2478/raon-2019-0055. PMID 31747379
- [Background] Alba JR, Basterra J, Ferrer JC, Santonja F, Zapater E. Hypothyroidism in patients treated with radiotherapy for head and neck carcinoma: standardised long-term follow-up study. J Laryngol Otol. 2016 May;130(5):478-81. doi: 10.1017/S0022215116000967. Epub 2016 Mar 15. PMID 26975210
- [Background] Massimino M, Gandola L, Collini P, Seregni E, Marchiano A, Serra A, Pignoli E, Spreafico F, Pallotti F, Terenziani M, Biassoni V, Bombardieri E, Fossati-Bellani F. Thyroid-stimulating hormone suppression for protection against hypothyroidism due to craniospinal irradiation for childhood medulloblastoma/primitive neuroectodermal tumor. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):404-10. doi: 10.1016/j.ijrobp.2007.03.028. Epub 2007 Jul 2. PMID 17601681
- [Background] Massimino M, Gandola L, Pignoli E, Seregni E, Marchiano A, Pecori E, Catania S, Cefalo G. TSH suppression as a possible means of protection against hypothyroidism after irradiation for childhood Hodgkins lymphoma. Pediatr Blood Cancer. 2011 Jul 15;57(1):166-8. doi: 10.1002/pbc.22915. Epub 2011 Feb 9. PMID 21557462
- [Background] Massimino M, Podda M, Gandola L, Pignoli E, Seregni E, Morosi C, Spreafico F, Ferrari A, Pecori E, Terenziani M. Long-term results of suppressing thyroid-stimulating hormone during radiotherapy to prevent primary hypothyroidism in medulloblastoma/PNET and Hodgkin lymphoma: a prospective cohort study. Front Med. 2021 Feb;15(1):101-107. doi: 10.1007/s11684-020-0752-2. Epub 2020 Aug 13. PMID 32794013
- [Background] Groover TA, Christie AC, Merritt EA, Coe FO, McPeak EM. Roentgen irradiation in the treatment of hyperthyroidism: a statistical evaluation based on three hundred and five cases. JAMA 1929; 92:1730-1734.
- [Background] Bantle JP, Lee CK, Levitt SH. Thyroxine administration during radiation therapy to the neck does not prevent subsequent thyroid dysfunction. Int J Radiat Oncol Biol Phys. 1985 Nov;11(11):1999-2002. doi: 10.1016/0360-3016(85)90283-4. PMID 3932271